CLINICAL TRIAL: NCT07245121
Title: Perineural Prolotherapy in Chronic Knee Osteoarthritis Pain: A Randomized Controlled Trial.
Brief Title: Perineural Prolotherapy in Chronic Knee Osteoarthritis Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Kalimeris, Associate Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 610/05-09-2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Perineural Analgesia; Prolotherapy; Knee Osteoarthritis
Keywords: Perineural prolotherapy; Knee osteoarthritis; Chronic pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextrose + Lidocaine group (group D+L) (Active Comparator): In the Dextrose + Lidocaine group (group D+L) an ultrasound guided perineural injection of DW 5% and lidocaine 1% will be performed at the 4 genicular nerves (superomedial, superolateral, inferomedial, recurrent peroneal genicular nerve).
  Interventions: Drug: Dextrose 5% and Lidocaine
- Lidocaine group (group L) (Active Comparator): In the lidocaine group (group L) an ultrasound guided perineural injection of a solution of lidocaine 1% will be performed at the 4 genicular nerves (superomedial, superolateral, inferomedial, recurrent peroneal genicular nerve).
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Dextrose 5% and Lidocaine — In the Dextrose + Lidocaine group (group D+L) a perineural infusion of a total volume of 8 ml of DW 5% and lidocaine 1% will be performed at the 4 genicular nerves (2ml per nerve), which will be prepared as follows: 4 ml of lidocaine 2%, with 1.2 ml of DW 35% and 2.8 ml of NaCl 0.9%. All perineural injections will be executed under ultrasound guidance 3 times (in 3 consecutive sessions): at their first assessment, 2 and 4 weeks later.
  Arms: Dextrose + Lidocaine group (group D+L)
Drug: Lidocaine — In the Lidocaine group (group L) the respective infusion of a solution of 8 ml of lidocaine 1% at the 4 genicular nerves (2ml per nerve) will be prepared as follows: 4 ml of lidocaine 2% with 4 ml of NaCl 0.9%. The perineural injections in each group will be executed 3 times (in 3 consecutive sessions): at their first assessment, 2 and 4 weeks later.
  Arms: Lidocaine group (group L)

SUMMARY:
The aim of this study is to test whether the addition of dextrose to perineural injections is superior to local anesthetic alone, as some initial data have indicated. To enhance the potential therapeutic effect, we will proceed to a 4-point injection technique, targeting 4 genicular nerves (superomedial, superolateral, inferomedial, recurrent peroneal genicular nerve) in a randomized controlled trial with two arms.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a common musculoskeletal disorder characterized by pain, stiffness, and decreased function of the affected joint. Based on the severity of the disease, the therapeutic approach can be either conservative - minimally invasive, or surgical. One of the implemented conservative methods is the desensitization of the genicular nerves, via perineural injection of local anesthetic, as they provide sensory innervation to the knee joint and participate in the pathophysiology of neuropathic pain of KOA. Ultrasound guidance has significantly improved the precision of local anesthetic injections, thereby enhancing the effectiveness of therapeutic interventions targeting these nerves. Since the genicular nerves are very small, injections are often performed close to the genicular arteries, which are more easily identified with ultrasound. The documented limited therapeutic effect of this approach and the complications of neurodestructive techniques, like thermal radiofrequencies, necessitate the use of alternative methods for the treatment of chronic pain in KOA.

Prolotherapy was introduced as a regenerative treatment involving the injection of a glucose solution into or around the joint space to stimulate repair and promote functional restoration of the joint's soft tissues. Perineural prolotherapy (glucose concentration DW 5%) seems to exert therapeutic effects by inhibiting the activation of the TRPV1 pain receptor located at the terminals of nociceptive neurons, thereby reducing the neurogenic inflammation and destruction of surrounding tissues. Also, separating the nerve through the non-specific mechanical effect of fluid under force (hydrodissection) gradually reduce adhesions, enhance blood flow, and mobilize the nerve to promote neuroregeneration. However, these data were derived from studies regarding nerve entrapment, but not for anatomically intact nerves like KOA, while there is no direct evaluation of perineural prolotherapy until today in knee pain.

The purpose of this clinical study is to test the hypothesis that perineural injection of 5% dextrose and lidocaine into 4 genicular nerves (superomedial, superolateral, inferomedial, recurrent peroneal genicular nerve) is superior to lidocaine injection in the treatment of chronic pain in patients with KOA.

Sample size calculation is for the primary outcome measure (i.e. pain score 15 days after the 3rd injection). Based on bibliographic data of similar studies (Fu Y et al 2024) was found that the Pain score (VAS) of patients treated with peri-articular perineural injection (PG) was 4.80 ± 1.005 while from the work of Kim et al 2018 was found that the VAS score for patients injected with lidocaine alone was 40.4 ± 9.1 which was converted to10 scale (4.04±0.91). Based on this is expected an effect size equal to 0.79. Furthermore, by study design is expected equal patient allocation in the two arms, in addition we considered error probability 5%, study power 80% and two tailed tests. The total sample size based on the previous data is 52 patients (equally allocated in two arms), and in order to compensate for possible dropouts we will enroll 60 patients.

After sample of 60 patients (30 patients in each group) will be enrolled in the prospective, randomized, single-blind, superiority, controlled, clinical trial. After patients written informed consent, they will be randomized with allocation ratio 1:1 to either dextrose + lidocaine group (intervention group) or lidocaine group (active control group). Randomization will be performed using computer-generated sequences to ensure allocation concealment, minimizing selection bias. Participants will be blinded to group assignment, whereas clinicians administering the injections will not be blinded due to the nature of the intervention. This single-blind approach balances methodological rigor with practical feasibility. Before the perineural injections in both groups, the pain intensity and its impact on daily life, including general activity, mood, sleep and social interactions will be evaluated via the self-report questionnaire <Brief Pain Inventory> (BPI), followed by the calculation of the Pain Severity and Pain Interference Score. In addition, the physical function of patients will be assessed via the 30 seconds chair stand test and the severity of knee osteoarthritis will be estimated via the questionnaire <Western Ontario and McMaster Universities arthritis index (WOMAC)> and the respective score will be subsequently calculated.

Procedure:

No oral or intravenous medication will be administered at the beginning or during the procedure. The patients' vital signs will be monitored during the procedure and appropriate sterilized conditions will be ensured. The locations for the infiltration of the 5 genicular nerves will be firstly identified after ultrasound examination and the subsequent ultrasound-guided perineural injection will be accomplished.

In the Dextrose + Lidocaine group (group D+L) a perineural infusion of a total volume of 8 ml of DW 5% and lidocaine 1% will be performed at the 4 genicular nerves, which will be prepared as follows: 4 ml of lidocaine 2%, with 1.2 ml of DW 35% and 2.8 ml of NaCl 0.9%. In the Lidocaine group (group L) the respective infusion of a solution of 8 ml of lidocaine 1% at the 4 genicular nerves will be prepared as follows: 4 ml of lidocaine 2% with 4 ml of NaCl 0.9%. The perineural injections in each group will be executed 3 times (in 3 consecutive sessions): at their first assessment, 2 and 4 weeks later.

Measurements

* Pain Severity Score at 15 days after the 3rd infiltration. It is one of the two main components of Brief Pain Inventory (BPI) score, a numerical scale used to assess pain. The Severity Score is an average of pain intensity ratings (worst, least, average, and current pain). Patients rate their pain on a 0-10 scale, with 0 being "no pain and 10 being "pain as bad as you can imagine".
* Pain Severity Score at baseline, 30 and 90 days after the 3rd infiltration. It will be estimated by the Brief Pain Inventory (BPI) score, as described above.
* Pain Interference Score at baseline, 15, 30 and 90 days after the 3rd infiltration. It is a main component of the Brief Pain Inventory (BPI) score, based on how pain affects daily life. Patients rate the impact of pain on life domains (like mood, sleep, and activities) on a 0-10 scale, with 0 being "no interference" and 10 being "completely interferes".
* Short-term changes 24h after the first infiltration. Approximately 24 hours after the 1st infiltration, a brief patient evaluation will be conducted. Specifically, pain intensity at the affected knee during movement will be assessed, according to Numerical Rating Scale (NRS), where patients assign a number from 0 to 10 to describe their pain level, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable". Furthermore, the duration of the analgesia provided by the perineural injection will be recorded, along with the patient's level of optimism regarding the treatment's effectiveness and its impact on improving daily life.
* WOMAC Questionnaire. Patients physical function will be evaluated by WOMAC questionnaire, which is divided into three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). The 24-item questionnaire uses a 0-4 scale (None to Extreme), where scores are summed for each subscale (Pain 0-20, Stiffness 0-8, Function 0-68). Higher WOMAC scores indicate worse symptoms and greater functional limitations. Measurement will be made at: baseline, 30 and 90 days after completion of the therapy. Further subitems of WOMAC questionnaire might also be evaluated.
* 30 seconds chair stand test (30CST). The number of successful attempts to stand up from a chair approximately 43 cm high, with a straight back and no arms for 30 seconds will be measured. Measurement will be made at: Baseline, 15, 30 and 90 days after completion of the therapy.
* Global Impression of Change (GIC) scale, a subjective patient rating of overall improvement after treatment. It will be documented at 90 days after the 3rd infiltration.
* Sub analyses of the scales used. Sub analyses of questions, eg. usage of analgesics.

Finally, any adverse events will be recorded.

STATISTICAL ANALYSIS Descriptive characteristics for the quantitative data will be expressed as median and Quartile 1 (Q1) to Quartile 3 (Q3), range or mean±standard deviation (SD) depending on normality as this will be checked by the Shapiro Wilk test. For the qualitative data will be reported the frequency of occurrence and the relevant percentage. Comparisons between the two arms at 15 days, depending on normality will be performed via the Mann Whitney U test or t-test. The significance level will be set to 0.05, and when applicable tests were two sided.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes
2. Age >38 years
3. Body Mass Index (BMI) up to 42 kg/m2
4. Diagnosis of knee osteoarthritis, according to the clinical criteria of the American College of Rheumatology. Osteoarthritis if the following combinations are present:

   A, B, C, D or A, B, E or A, D, E:

   A) Knee pain most days of the previous month B) Cracking during active joint movement C) Morning stiffness lasting at least 30 minutes D) Age at least 38 years E) Bone swelling of the affected knee on physical examination
5. Chronic knee pain on the Numerical Rating Scale (NRS) > 5 for at least 3 months prior to the study
6. Grade 2 or 3 osteoarthritis, according to the Kellgern-Lawrence classification
7. Pain, creaking, and stiffness in the knee joint that persists for at least three months prior to the study.

Exclusion Criteria:

1. Any infection of the skin of the knee joint, such as cellulitis, or periarticular or intraarticular infection during the last 3 months
2. Poorly controlled diabetes mellitus or connective tissue disease affecting the knee joint
3. History of previous total knee arthroplasty or other knee surgery.
4. History of periarticular or intraarticular injection of corticosteroids, local anesthetic, hyaluronic acid, platelet-rich plasma, radiofrequency, prolotherapy within the last trimester
5. History of knee injury or fracture within the last 3 months
6. History of acute lumbosacral radiculopathy or peripheral neuropathy, neurological, psychiatric disease
7. Pain limited in the posterior aspect of the knee
8. History of limb malignancy
9. History of bleeding disorder
10. Pregnancy
11. Allergy to local anesthetics, needle phobia
12. Difficulty communicating (severe hearing loss, dementia, language problems)
13. Non-guaranteed transportation to hospital for treatments and re-evaluations

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pain Severity Score (PSS) at 15 days after the 3rd (last) infiltration | 15 days after the 3rd infiltration of the first participant up to 15 days after the 3rd infiltration of the last participant
  The primary outcome will be estimated by the Brief Pain Inventory (BPI) score, a numerical scale used to assess pain. This score is the arithmetic average of four items related to pain intensity: worst pain, least pain, average pain, and current pain (SCORE RANGE: 0= No pain, 1-3= Mild pain, 4-6= Moderate pain, 7-10= Severe pain).

SECONDARY OUTCOMES:
Pain Severity Score (PSS) at baseline, 30 and 90 days after the 3rd infiltration | A measurement before the first infiltration of the first participant up to 90 days after the 3rd infiltration of the last participant.
  It will be estimated by the Brief Pain Inventory (BPI) score. This score is the arithmetic average of four items related to pain intensity: worst pain, least pain, average pain, and current pain (SCORE RANGE: 0= No pain, 1-3= Mild pain, 4-6= Moderate pain, 7-10= Severe pain).
Pain Interference Score (PIS) | From before the first infiltration of the first participant up to 3 months after the last infiltration of the last participant.
  Pain Interference Score from the relevant items of the Brief Pain Inventory (BPI) Score at baseline, 15, 30 and 90 days after the last infiltration. This score is the arithmetic average of seven items that assess how pain interferes with daily functions: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life (SCORE RANGE: 0= No interference, 1-3= Mild interference, 4-6= Moderate interference, 7-10= Severe interference).
Short-term changes 24h after the first infiltration | 24 hours after the first infiltration of the first participant up to 24 hours after the first infiltration of the last participant.
  Pain intensity at the affected knee during movement will be assessed, according to Numerical Rating Scale (NRS), where patients assign a number from 0 to 10 to describe their pain level, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable". Furthermore, the duration of the analgesia provided by the perineural injection will be recorded, along with the patient's level of optimism regarding the treatment's effectiveness and its impact on improving daily life.
WOMAC Questionnaire | Baseline, 15, 30 and 90 days after completion of the therapy of the first participant until 90 days after completion of therapy of the last participant.
  Patients physical function will be evaluated by WOMAC questionnaire, which is divided into three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). The 24-item questionnaire uses a 0-4 scale (None to Extreme), where scores are summed for each subscale (Pain 0-20, Stiffness 0-8, Function 0-68). Higher WOMAC scores indicate worse symptoms and greater functional limitations. Measurement will be made at: baseline, 15, 30 and 90 days after completion of the therapy. Further subitems of WOMAC questionnaire might also be evaluated.
30 seconds chair stand test (30CST) | Baseline, 15, 30 and 90 days after completion of the therapy of the first participant until 90 days after completion of therapy of the last participant.
  30 seconds chair stand test, where the number of successful attempts to stand up from a chair approximately 43 cm high, with a straight back and no arms for 30 seconds will be measured.
  Measurement will be made at: Baseline, 15, 30 and 90 days after completion of the therapy.
The Global Impression of Change (GIC) scale | 3 months after completion of therapy for the first participant up to 3 months after completion of therapy for the last participant.
  Score according to the Global Impression of Change (GIC) scale (a subjective patient rating of overall improvement after treatment). It will be documented at 90 days after the 3rd infiltration.

OTHER OUTCOMES:
Subanalyses of the scales used | Baseline, 15, 30 and 90 days after completion of the therapy of the first participant until 90 days after completion of therapy of the last participant
  Subanalyses of questions, eg. usage of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kalimeris, Assoc Prof of Anesthesiology, Study Chair — National and Kapodistrian University of Athens; Theodosios Saranteas, Professor of Anesthesiology, Study Chair — National and Kapodistrian University of Athens; Andreas Maurogenis, Assoc Prof of Anesthesiology, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- University General Hospital of Athens "Attikon" - National and Kapodistrian University of Athens Medical School, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim DH, Choi SS, Yoon SH, Lee SH, Seo DK, Lee IG, Choi WJ, Shin JW. Ultrasound-Guided Genicular Nerve Block for Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial of Local Anesthetic Alone or in Combination with Corticosteroid. Pain Physician. 2018 Jan;21(1):41-52. PMID 29357330
- [Background] Ahmed A, Arora D. Ultrasound-guided radiofrequency ablation of genicular nerves of knee for relief of intractable pain from knee osteoarthritis: a case series. Br J Pain. 2018 Aug;12(3):145-154. doi: 10.1177/2049463717730433. Epub 2017 Sep 19. PMID 30057759
- [Background] Waluyo Y, Artika SR, Insani Nanda Wahyuni, Gunawan AMAK, Zainal ATF. Efficacy of Prolotherapy for Osteoarthritis: A Systematic Review. J Rehabil Med. 2023 Feb 27;55:jrm00372. doi: 10.2340/jrm.v55.2572. PMID 36847731
- [Background] Farpour HR, Fereydooni F. Comparative effectiveness of intra-articular prolotherapy versus peri-articular prolotherapy on pain reduction and improving function in patients with knee osteoarthritis: A randomized clinical trial. Electron Physician. 2017 Nov 25;9(11):5663-5669. doi: 10.19082/5663. eCollection 2017 Nov. PMID 29403602
- [Background] Rabago D, Patterson JJ, Mundt M, Kijowski R, Grettie J, Segal NA, Zgierska A. Dextrose prolotherapy for knee osteoarthritis: a randomized controlled trial. Ann Fam Med. 2013 May-Jun;11(3):229-37. doi: 10.1370/afm.1504. PMID 23690322
- [Background] Rezasoltani Z, Taheri M, Mofrad MK, Mohajerani SA. Periarticular dextrose prolotherapy instead of intra-articular injection for pain and functional improvement in knee osteoarthritis. J Pain Res. 2017 May 17;10:1179-1187. doi: 10.2147/JPR.S127633. eCollection 2017. PMID 28553139
- [Background] Ebnerasooli S, Barghi A, Nasseri K, Moghimi N. Peri-articular Dextrose Prolotherapy: Investigating the Effect of Injection Site on Knee Osteoarthritis Pain: A Double-Blind, Randomized, Clinical Trial. Anesth Pain Med. 2024 Mar 27;14(2):e140966. doi: 10.5812/aapm-140966. eCollection 2024 Apr. PMID 39411379
- [Background] Ghai B, Kumar M, Makkar JK, Goni V. Comparison of ultrasound guided pulsed radiofrequency of genicular nerve with local anesthetic and steroid block for management of osteoarthritis knee pain. Korean J Pain. 2022 Apr 1;35(2):183-190. doi: 10.3344/kjp.2022.35.2.183. PMID 35354681
- [Background] Chen JL, Chen CH, Cheng CH, Chen CC, Lin KY, Chen CPC. Can the addition of ultrasound-guided genicular nerve block using 5% dextrose water augment the effect of autologous platelet rich plasma in treating elderly patients with knee osteoarthritis? Biomed J. 2021 Dec;44(6 Suppl 1):S144-S153. doi: 10.1016/j.bj.2020.08.011. Epub 2020 Sep 1. PMID 35289285
- [Background] Fu Y, Du Y, Li J, Xi Y, Ji W, Li T. Demonstrating the effectiveness of intra-articular prolotherapy combined with peri-articular perineural injection in knee osteoarthritis: a randomized controlled trial. J Orthop Surg Res. 2024 May 5;19(1):279. doi: 10.1186/s13018-024-04762-4. PMID 38705988
- [Background] Bhargava M, Gaur R, Gonnade NM, Sarankumar G, Elhence A, Gahlot N. Comparing effectiveness of 3-needle approach versus 5-needle approach of genicular nerve block on pain and quality of life in chronic osteoarthritis of knee: a double blinded randomised controlled trial. BMC Musculoskelet Disord. 2024 Nov 29;25(1):978. doi: 10.1186/s12891-024-07938-5. PMID 39614201
- [Background] Govender-Davies S, Davies L, Pillay-Addinall S. A cadaveric study investigating the spread of injectate following an interspace between the popliteal artery and the capsule of the posterior knee block in a neonatal sample: a pilot study. Anat Cell Biol. 2024 Jun 30;57(2):229-237. doi: 10.5115/acb.23.274. Epub 2024 Mar 29. PMID 38551026
- [Background] Yin W, Luo D, Xu W, Yang W, Jia S, Lin J. Effect of adductor canal block combined with infiltration between the popliteal artery and posterior capsular of the knee on chronic pain after total knee arthroplasty: a prospective, randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2024 Sep 10;24(1):320. doi: 10.1186/s12871-024-02707-2. PMID 39256652
- [Background] Wu YT, Chen YP, Lam KHS, Reeves KD, Lin JA, Kuo CY. Mechanism of Glucose Water as a Neural Injection: A Perspective on Neuroinflammation. Life (Basel). 2022 Jun 2;12(6):832. doi: 10.3390/life12060832. PMID 35743863
- [Background] Kim H, Kim HJ, Jung YH, Do W, Kim EJ. The effect of perineural injection therapy on neuropathic pain: a retrospective study. J Dent Anesth Pain Med. 2024 Feb;24(1):47-56. doi: 10.17245/jdapm.2024.24.1.47. Epub 2024 Feb 1. PMID 38362256
- [Background] Yildirim Uslu E. Ultrasound-Guided Perineural Dextrose Injection for Superior Cluneal Nerve Neuropathy Treatment. Cureus. 2024 Sep 26;16(9):e70229. doi: 10.7759/cureus.70229. eCollection 2024 Sep. PMID 39463523